CLINICAL TRIAL: NCT03778294
Title: Phase II Study of Short Course Hypofractionated Proton Beam Therapy Incorporating 18F-DOPA-PET/MRI for Elderly Patients With Newly Diagnosed Glioblastoma
Brief Title: 18F-DOPA-PET/MRI Scan in Imaging Elderly Patients With Newly Diagnosed Grade IV Malignant Glioma or Glioblastoma During Planning for a Short Course of Proton Beam Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1774; NCI-2018-02800 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1774 (Other: Mayo Clinic); 17-007458 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2023-12

CONDITIONS: Glioblastoma; Malignant Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — fluorodopa F 18; Magnetic Resonance Spectroscopy; Proton Therapy; Protons; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (18F-DOPA, PET/MRI, PET/CT, temozolomide) (Experimental): Patients receive 18F-DOPA IV and undergo PET/MRI or PET/CT imaging scan. Patients then receive proton beam radiotherapy over 5 or 10 consecutive days excluding weekend and standard of care temozolomide on days 1-7 or 1-14. Beginning cycles 2, patients receive standard of care temozolomide on days 1-5. Cycles with temozolomide repeat every 28 days for up to 7 cycles in the in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Computed Tomography; Other: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fluorodopa F 18 — Given IV
  Other Names: (18F)FDOPA; 18F-DOPA; 18F-FDOPA; 3-(2-Fluoro-(sup 18)F-4,5-dihydroxyphenyl)-L-alanine; 6-(18F)Fluoro-L-DOPA; Fluorine F 18 Fluorodopa; Fluorine-18-fluoro-L-DOPA; Fluorodopa (18F); FLUORODOPA F-18; L-6-(18F)Fluoro-DOPA
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Proton Beam Radiation Therapy — Receive proton beam RT
  Other Names: PBRT; Proton; Proton Radiation Therapy; Radiation, Proton Beam
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Temozolomide — Drug
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies how well fluorodopa F 18-positron emission tomography/magnetic resonance imaging scan (18F-DOPA-PET/MRI) works in imaging elderly patients with newly diagnosed grade IV malignant glioma or glioblastoma during planning for a short course of proton beam radiation therapy. 18F-DOPA is a chemical tracer that highlights certain cells during imaging. PET scan, is a metabolic imaging technique which takes advantage of how tumor cells take up nutrients differently than normal tissue. MRI scans are used to guide radiation therapy for most brain tumors. Hypofractionated proton beam therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Using 18FDOPA-PET scans along with MRI scans may be able to provide the radiation doctor with information on tumor tissue versus normal, healthy tissue and may help the doctor more accurately plan the radiation treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare overall survival at 12 months for grade IV glioma patients after radiation therapy targeting volumes designed with both 18F-DOPA-PET and conventional magnetic resonance (MR) image (or PET/computed tomography [CT]) information with historical controls.

SECONDARY OBJECTIVES:

I. Compare progression free survival at 12 months after radiation therapy targeting volumes designed with both 18F-DOPA-PET and conventional MR image information with historical controls.

II. Determine acute and late effect toxicity after hypofractionated proton beam radiotherapy treatment including areas of high 18F-DOPA-PET uptake (T/N > 2.0).

CORRELATIVE RESEARCH OBJECTIVES:

I. Compare radiotherapy (RT) treatment volumes defined by MR only with RT treatment volumes defined with both PET and MR information for grade IV glioma patients.

II. Compare differences in RT volumes identified using biopsy-validated thresholds as highly aggressive disease comparing 18F-DOPA uptake and relative cerebral blood volume (relCBV) from perfusion MRI (pMRI) as well as differences in RT volumes identified using biopsy-validated thresholds as tumor extent comparing 18F-DOPA uptake and diffusion maps from diffusion tensor imaging (DTI) will be evaluated.

III. Evaluate quality of life after radiotherapy using European Organization for Research and Treatment of Cancer (EORTC) questionnaires compared with historical controls from Keim-Guibert et al.

IV. Compare differences in proton radiation planning utilizing radiobiologic modeling/evaluation techniques performed at Mayo Clinic Rochester to linear energy transfer distribution evaluation at Mayo Clinic Arizona.

OUTLINE:

Patients receive 18F-DOPA intravenously (IV) and undergo PET/MRI or PET/CT imaging scan. Patients then receive proton beam radiotherapy over 5 or 10 consecutive days excluding weekend and standard of care temozolomide on days 1-7 or 1-14. Beginning cycles 2, patients receive standard of care temozolomide on days 1-5. Cycles with temozolomide repeat every 28 days for up to 7 cycles in the in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 1 year, and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed grade IV malignant glioma
* Planned radiation treatments at Mayo Clinic Arizona or Mayo Clinic Rochester
* Willing to sign release of information for any radiation and/or follow-up records
* Provide informed written consent
* Patients with estimated glomerular filtration rate (eGFR) >= 60 mg/min/1.72 m^2
* Ability to complete questionnaire(s) by themselves or with assistance
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2

Exclusion Criteria:

* Patients diagnosed with grades I-III glioma
* Currently on Avastin at time of treatment
* Unable to undergo MRI scans with contrast (e.g. cardiac pacemaker, defibrillator, kidney failure)
* Unable to undergo an 18F-DOPA-PET scan (e.g. Parkinson's disease, taking anti-dopaminergic, or dopamine agonist medication or less than 6 half-lives from discontinuance of dopamine agonists)

  * NOTE: Other potentially interfering drugs: amoxapine, amphetamine, benztropine, buproprion, buspirone, cocaine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, selegiline, paroxetine, citalopram, and sertraline. If a patient is on any of these drugs, list which ones on the on-study form
* Pregnant women, nursing women, or men or women of childbearing potential who are unwilling to employ adequate contraception.

  * NOTE: All women enrolled in this study will be age 65 or over, and at the determination of the principal investigator (PI), will not be of childbearing potential. If the radiology department requires a pregnancy test before administering the 18FDOPA injection, they may perform one per their standard of care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sujay A Vora, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Vora S, Pafundi D, Voss M, Buras M, Ashman J, Bendok B, Breen W, Hu L, Kizilbash S, Laack N, Liu W, Mahajan A, Mrugala M, Porter A, Ruff M, Sio T, Uhm J, Yang M, Brinkmann D, Brown P. Short-course hypofractionated proton beam therapy, incorporating 18F-DOPA PET and contrast-enhanced MRI targeting, for patients aged 65 years and older with newly diagnosed glioblastoma: a single-arm phase 2 trial. Lancet Oncol. 2024 Dec;25(12):1625-1634. doi: 10.1016/S1470-2045(24)00585-0. Epub 2024 Nov 18. PMID 39571596

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide): Patients receive 18F-DOPA IV and undergo PET/MRI or PET/CT imaging scan. Patients then receive proton beam radiotherapy over 5 or 10 consecutive days excluding weekend and standard of care temozolomide on days 1-7 or 1-14. Beginning cycles 2, patients receive standard of care temozolomide on days 1-5. Cycles with temozolomide repeat every 28 days for up to 7 cycles in the in the absence of disease progression or unacceptable toxicity.> > Computed Tomography: Undergo PET/CT>
  > Fluorodopa F 18: Given IV>
  > Magnetic Resonance Imaging: Undergo PET/MRI>
  > Positron Emission Tomography: Undergo PET/CT or PET/MRI>
  > Proton Beam Radiation Therapy: Receive proton beam RT>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies>
  > Temozolomide: Drug
Period: Overall Study
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
Started | 43
Completed | 39
Not Completed | 4
Not completed — Death | 1
Not completed — Issues with insurance | 1
Not completed — disease progression before treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.617 (5.097)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 37
  More than one race | 0
  Unknown or Not Reported | 1
Corticosteroid therapy at study entry? [Count of Participants; unit: Participants]
  Yes | 21
  No | 18
Path result/Molecular factors [Count of Participants; unit: Participants]
  IDH1 mutant | 0
  IDH1 Wildtype | 39
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction. > ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. > ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. > ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 13
    1 | 19
    2 | 7
Neurological Deficit [Count of Participants; unit: Participants]
  Yes | 13
  No | 26
History of seizure [Count of Participants; unit: Participants]
  Yes | 10
  No | 29
Extent of surgery [Count of Participants; unit: Participants]
  Gross total resection | 16
  Subtotal resection | 8
  Biopsy | 15
MGMT [Count of Participants; unit: Participants]
  Methylated | 13
  Unmethylated | 24
  Not available | 2
Family history of brain tumor [Count of Participants; unit: Participants]
  Yes | 1
  No | 38
Use of alternating electrical therapy [Count of Participants; unit: Participants]
  Yes | 0
  No | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated utilizing exact binomial methodology. The distribution of survival time will be estimated using the method of Kaplan-Meier (1958).
Time Frame: Time from registration to death due to any cause, assessed up to 12 months
Measure: Number (90% Confidence Interval); unit: proportion of successes
Groups:
- Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide): Patients receive 18F-DOPA IV and undergo PET/MRI or PET/CT imaging scan. Patients then receive proton beam radiotherapy over 5 or 10 consecutive days excluding weekend and standard of care temozolomide on days 1-7 or 1-14. Beginning cycles 2, patients receive standard of care temozolomide on days 1-5. Cycles with temozolomide repeat every 28 days for up to 7 cycles in the in the absence of disease progression or unacceptable toxicity.
  >
  > Computed Tomography: Undergo PET/CT
  >
  > Fluorodopa F 18: Given IV
  >
  > Magnetic Resonance Imaging: Undergo PET/MRI
  >
  > Positron Emission Tomography: Undergo PET/CT or PET/MRI
  >
  > Proton Beam Radiation Therapy: Receive proton beam RT
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
  >
  > Temozolomide: Drug
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
Number analyzed (Participants) | 39
proportion of successes | 0.54 [0.43 to 1.0]

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from registration to the earliest date documenting disease progression
Time Frame: At 12 months after radiation therapy
Measure: Number (95% Confidence Interval); unit: proportion of successes
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
Number analyzed (Participants) | 39
proportion of successes | 0.72 [0.55 to 0.85]

3. Secondary Outcome: Progression Free Survival
Description: Defined as the time from registration to the earliest date documenting disease progression
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
Number analyzed (Participants) | 39
months | 6.9 [6.01 to 9.66]

4. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The rate of acute and late treatment-related toxicities for newly diagnosed high-grade glioma patients treated with fluorodopa F 18-positron emission tomography (18F-DOPA PET) image-guided hypofractionated proton beam therapy will be determined, with acute radiotherapy (RT) toxicities graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
Number analyzed (Participants) | 39
Participants
  Grade 2 Post Baseline | 34
  Grade 3 Post Baseline | 18
  Grade 4 Post Baseline | 5
  Grade 2 Acute | 27
  Grade 3 Acute | 7
  Grade 4 Acute | 0
  Grade 2 Late | 24
  Grade 3 Late | 14
  Grade 4 Late | 5

5. Other Pre Specified Outcome: Radiotherapy (RT) Treatment Volumes
Description: Paired t-test statistical analysis will be performed to determine if any differences exist and the level of statistical significance between treatment volumes defined by magnetic resonance (MR) only and treatment volumes defined with both positron emission tomography (PET) and MR information.
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Quality of Life (QOL)
Description: QOL surveys will be compared to data from historical controls. Quality of life will be assessed at baseline and at each magnetic resonance imaging (MRI) evaluation (up to 6 evaluations). QOL will be measured using the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30, a 30-item patient-reported questionnaire about patient ability to function, symptoms related to the cancer and its treatment, overall health and quality of life, and perceived financial impact of the cancer and its treatment. 28 of the 30 items are measured on a 1-4 scale (1=not at all; 4=very much) with the remaining two items (overall health and overall quality of life) scored on a 1-7 numeric analogue scale (1=very poor; 7=excellent). The recall period for the EORTC QLQ-C30 is one week. Higher scores indicate better QoL for overall health status and functioning scales, and worse QoL for symptom scales
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Differences in Proton Radiation Planning
Description: Paired t-test statistical analysis will be performed to determine if any differences exist and the level of statistical significance between proton plan metrics based off two modeling/evaluation techniques: radiobiologic modeling/evaluation techniques performed at Mayo Clinic Rochester and Linear Energy Transfer (LET) distribution evaluation at Mayo Clinic Arizona
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide)
All-Cause Mortality (participants affected / at risk) | 32/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 39/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (18F-DOPA, PET/MRI, PET/CT, Temozolomide) (N=39)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 36 (135)
Pain (General disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Lymphocyte count decreased (Investigations) | 11 (18)
Platelet count decreased (Investigations) | 9 (10)
Weight loss (Investigations) | 8 (16)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 24 (48)
Concentration impairment (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 4 (4)
Encephalopathy (Nervous system disorders) | 11 (14)
Headache (Nervous system disorders) | 21 (40)
Memory impairment (Nervous system disorders) | 3 (3)
Muscle weakness left-sided (Nervous system disorders) | 2 (7)
Muscle weakness right-sided (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 16 (21)
Agitation (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 20 (41)
Irritability (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (71)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03778294/Prot_SAP_000.pdf